CLINICAL TRIAL: NCT07224464
Title: Open Label Feasibility Dose Escalation Study to Evaluate the Safety of Sarah Nanotechnology System, With Alternating Magnetic Field (AMF) Application in Patients With Advanced Metastatic Solid Tumors.
Brief Title: The Sarah Nanotechnology System for Treatment of Advanced Metastatic Solid Tumors Using Hyperthermia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Phase Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL-400-001
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Solid Tumors; Stage 4 Cancer
Keywords: Advanced metastatic solid tumors; Stage 4 cancer; Stage 4 liver cancer; Stage 4 ovarian cancer; Stage 4 colon cancer; Stage 4 breast cancer; Stage 4 lung cancer; Stage 4 cervical cancer; Stage 4 cholangiocarcinoma; Hyperthermia; Metastatic Solid Tumors
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lung Neoplasms; Uterine Cervical Neoplasms; Cholangiocarcinoma; Hyperthermia | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Level 1 (Experimental): 1.2 mg/kg of SaNP (Sarah nanoparticles) with 12-15 min of AMF irradiation
  Interventions: Device: The Sarah Nanotechnology System - intended to deliver thermal energy to malignant cells for the purpose of thermal destruction of these cells in patients with advanced metastatic solid tumors.
- Level 2 (Experimental): 1.2 mg/kg of SaNP (Sarah nanoparticles) with 16-20 min of AMF irradiation
  Interventions: Device: The Sarah Nanotechnology System - intended to deliver thermal energy to malignant cells for the purpose of thermal destruction of these cells in patients with advanced metastatic solid tumors.

INTERVENTIONS:
Device: The Sarah Nanotechnology System - intended to deliver thermal energy to malignant cells for the purpose of thermal destruction of these cells in patients with advanced metastatic solid tumors. — This intervention includes the use of intravenus injection of Sarah Nanoparticles (SaNP) containing iron oxide core, together with non-ionizing alternating magnetic field (AMF) radiation.
  Other Names: Hyperthermia

SUMMARY:
This is a sequential, dose-escalation, non-randomized, prospective, early feasibility trial. The goal of this clinical trial is to gather information on the safety and the recommended dose of the Sarah Nanotechnology System. Eligible participants have stage 4 metastatic solid tumor(s), that is(are) not responding to conventional treatment or have declined standard treatment options.

The main question it aims to answer is:

• What is the safety profile of the Sarah Nanotechnology System and which field strength and time of irradiation are safe for people?

Study participation involves:

* One intravenous injection (through a vein in the arm) of a solution that contains tiny particles (nanoparticles) containing iron oxide. The nanoparticles are delivered to the tumor(s) through blood circulation.
* About 4 hours after injection of the nanoparticles, participants are placed inside a machine (magnetic field system) where the upper torso will be exposed to low frequency (~300 kHz) alternating magnetic field (AMF) radiation. This type of radiation, unlike CT or X- rays, is non-ionizing. Non-ionizing means radiation that lacks the energy to remove electrons from an atom. Examples of devices that produce non-ionizing radiation are MRI machines, cell phones, Wi-Fi, microwave ovens, and sunlight.

The AMF heats up the iron oxide core in the nanoparticles, due to their magnetic properties, which in turn causes the temperature to increase within the tumor(s). Because cancer cells are more sensitive to heat than normal cells, the heat will damage the cancer cells potentially without harming the surrounding healthy tissues.

* During the treatment participants are covered by a cooling blanket to control body temperature, which will be monitored continuously throughout the procedure.
* Participants are followed up at 1 week and 1 month, and up to 5 years after the one-time treatment.

DETAILED DESCRIPTION:
This is a sequential, open-label, dose-escalation, non-randomized, prospective early feasibility clinical investigation designed to evaluate the safety of the Sarah Nanotechnology System, comprising intravenously administered Sarah Nanoparticles (SaNPs) in combination with a low-frequency Alternating Magnetic Field (AMF) generated by the Electromagnetic Induction System (EIS).

The purpose of the study is to assess the safety profile of the SaNP and AMF combination and to identify the recommended dose and irradiation parameters for a subsequent feasibility study. The study will also provide initial information regarding device performance and efficacy.

Scientific and Technical Background:

The Sarah Nanotechnology System utilizes controlled magnetic hyperthermia to thermally damage malignant cells while sparing surrounding healthy tissue. Following a single intravenous administration, SaNPs, nanoparticles with iron oxide core, circulate systemically and preferentially accumulate within tumor tissue through the Enhanced Permeability and Retention (EPR) effect, then participant's upper torso is exposed to an AMF (≈ 290 ± 10% kHz) by the EIS (Electromagnetic Induced System). The obtained effect is heating at tumor site.

Because AMF exposure can also induce eddy currents on the skin surface a patient cooling blanket system continuously helps regulating body surface temperature. Vital signs and skin temperature are monitored in real time throughout irradiation.

Dose-Escalation Design:

The study follows a standard 3 + 3 sequential escalation design, once the recommended dose is identified, an expansion cohort will repeat it.

SaNP dose: 100% SaNP dose, calculated according to NOAEL. AMF parameters: 290 ± 10% kHz; total irradiation time up to 15 minutes in the first treatment cohort, increasing to 16-20 minutes at the next treatment cohort depending on safety review.

Dose-limiting toxicity (DLT) criteria and escalation rules follow standard early-phase device study methodology.

Treatment Procedure:

On the treatment day, participants undergo laboratory tests and ECG assessment before SaNP infusion. Approximately four hours post-infusion, participants are positioned within the EIS coil for AMF irradiation while covered by a cooling blanket, and analgesic administration per physician discretion. Skin surface and oral temperatures, vital signs, and participant comfort are continuously monitored. After irradiation, repeat laboratory and ECG evaluations are performed prior to discharge.

Follow-up assessments occur at 7 ± 2 days and 30 ± 5 days post-treatment and then every 3-6 months up to 5 years for long-term safety surveillance.

Adverse events (AEs) and serious adverse events (SAEs) will be documented and evaluated for severity and relatedness to device or procedure. Real-time safety oversight is performed by the investigator and sponsor medical monitor; the DSMB periodically reviews cumulative safety data and recommends escalation, expansion, or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy of at least 90 days.
2. Histologically confirmed advanced metastatic solid tumors located between the thoracic inlet and the pelvic floor, that have progressed on or after standard therapy and are ineligible for surgical resection or local therapies.
3. Must have measurable disease according to RECIST 1.1.
4. Patient has exhausted all standard treatment options.
5. There must be resolution of all systemic treatment-related adverse events. At least 14 days must have elapsed since the last systemic or radiotherapy treatment before screening visit.
6. Documented progressive disease confirmed by either CT (chest and abdomen), MRI or PET/CT scan since patient's last cancer therapy.
7. No prior history of brain metastasis confirmed by CT or MRI within 30 days prior to treatment.
8. Treatment planning CT scan performed within 14 days prior to study treatment.
9. Age ≥18 years.
10. Rib cage circumference ≤ 90 cm.
11. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
12. Patients should have sufficient organ and bone marrow function on screening day and on procedure day as defined below:

    Leukocytes ≥3,000/mcL Absolute neutrophil count ≥1,500/mcL Platelets ≥100,000/mcL Total bilirubin ≤ 2.5 x limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤5 x institutional ULN Creatinine Glomerular filtration rate (GFR) ≥50 ml/min/1.73 m2 for patients with creatinine levels above institutional normal.
13. Ability to provide written informed consent document.
14. Confirmation that patient has no electronic or electronically conductive implants or metals:

    * Via a review of the CT scan
    * Metal questionnaire filled in by patients

Exclusion Criteria:

1. Received chemotherapy, radiotherapy or hormonal therapy within 14 days (before screening).
2. Received immunotherapy/biological therapy or any other investigational agent in the last 21 days (before screening).
3. Not yet recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1).
4. Presence of brain metastases or prior history of brain metastases (if no prior history, confirmed by CT or MRI within 30 days prior to treatment).
5. Known history of allergic reactions attributed to compounds of similar chemical or biological composition (For example: PEG 20,000 Dalton).
6. Uncontrolled intercurrent illness (including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, ischemia, or psychiatric illness) that in the opinion of the investigator would either limit compliance with study requirements or put participant at risk.
7. Pregnant and/or breastfeeding.
8. Unwilling to be abstinent or on contraception for up to 30 days after the last study treatment.
9. Presence of electronic or electronically conductive implants or metals in body (verified by screening CT and metal questionnaire).
10. Rib cage circumference over 90 cm.
11. Unable to provide written informed consent.
12. Unable to lay down with hands extended over head.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Primary safety profile: assessing the number of device related adverse events and serious adverse events. | From treatment day and up to 1 month post treatment.
  Evaluating the safety profile of the SaNP application via intravenous administration and the safety of the AMF radiation, in metastatic solid tumor patients, by assessing the procedural adverse events, and serious adverse events.
Primary safety of recommended dose: characterization of protocol dosing regimen | From treatment day and up to 1 month post treatment.
  Determining the recommended dose for the next efficacy study based on the different treatment arms.

SECONDARY OUTCOMES:
Secondary - Initial efficacy evaluation: assessing clinical response according to RECIST 1.1 | From treatment day and up to 1 month post treatment.
  Assessing response to treatment with SaNP and AMF radiation in participants with solid tumors according to evaluation, 1 month post treatment, of dynamic changes in the irradiated volume compared to baseline CT, using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Lester, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
This is an early feasibility study, the data is very preliminary as the sponsor (New Phase) is looking for the recommended treatment protocol for the next study.